CLINICAL TRIAL: NCT03423056
Title: Efficacy and Safety of a Preoperative Aerobic Exercise Program in Patients With Gastrointestinal Cancer. A Phase II Clinical Trial
Brief Title: Efficacy and Safety of a Preoperative Aerobic Exercise Program in Patients With Gastrointestinal Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Collaborators: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C41030617-091
Record Dates: First submitted 2018-01-11; First posted 2018-02-06 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-01

CONDITIONS: Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Liver Neoplasm
Keywords: Gastrointestinal Neoplasms; Exercise; Preoperative Period; Preoperative Care
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Liver Neoplasms; Gastrointestinal Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The individualized aerobic training program will be developed according to Karvonem's equation . It will programmed in 3 sessions/week (not in row) during 4 weeks
  Each 50-minutes session will be organized in three phases: warm up, central and back to calm. The heart rate target will be prescribed as follows:
  * Week 1: heart rate target: 50% of maximum heart rate
  * Week 2: heart rate target: 60% of maximum heart rate
  * Week 3: heart rate target: 70% of maximum heart rate
  * Week 4: heart rate target: 60% of maximum heart rate
  The aerobic exercise will be carried on a treadmill or in a stationary bicycle, according to the patient's preferences and will be supervised by a physical therapist.
  The post intervention aerobic capacity will be measured at week 3 and 4 with the 6-minute walk test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative exercise program (Experimental): The individualized aerobic training program will be developed according to Karvonem's equation . It will programmed in 3 sessions/week (not in row) during 4 weeks.
  Each 50-minutes session will be organized in three phases: warm up, central and back to calm. The heart rate target will be prescribed as follows:
  Week 1: heart rate target: 50% of maximum heart rate Week 2: heart rate target: 60% of maximum heart rate Week 3: heart rate target: 70% of maximum heart rate Week 4: heart rate target: 60% of maximum heart rate The aerobic exercise will be carried on a treadmill or in a stationary bicycle, according to the patient's preferences and will be supervised by a physical therapist.
  Interventions: Other: Preoperative exercise program

INTERVENTIONS:
Other: Preoperative exercise program — Individualized aerobic training program developed by physical therapist using Karvonem's equation . It will programmed in 3 sessions/week (not in row) during 4 weeks. Each 50-minutes session will be organized in three phases: warm up, central and back to calm. The heart rate target will be prescribed between 50 to 70% of the maximum heart rate and will be carried on a treadmill or in a stationary bicycle.
  Other Names: Preoperative aerobic exercise short program

SUMMARY:
Patients with gastrointestinal cancer often experience physical deconditioning; this could lead to an increased risk of complications, especially when they require major abdominal surgical procedures.

It has been suggested that physical training in the preoperative period could improve their condition, reducing the risk of complications. Although this topic has been investigated, it has not been established yet the best short preoperative aerobic exercise program to enhance the aerobic capacity in patients with gastrointestinal cancer who are going to be to surgical primary management, and consequently, to help patients dealing with the physiological stress involved in a surgical intervention.

Main objective:

To determine the efficacy and safety of a 4 weeks preoperative exercise program in patients with gastrointestinal cancer scheduled for primary surgery.

Materials and methods:

This is a Phase II single arm clinical trial that will include patients between 45 and 70 years, with confirmed gastrointestinal cancer (gastric, hepatic, colon or rectal cancer), without electrocardiographic abnormalities, and scheduled for primary surgery in 4 weeks or more since recruitment

All the enrolled patients will receive a basal aerobic capacity assessment with the 6-minute walk test. Then, two physical therapist will prescribe them a supervised and individualized aerobic training program in 3 sessions per week during 4 weeks. Each session will last 50 minutes and will increase the heart rate target weekly (from 50% to 70% of the maximum heart rate). The aerobic exercise will be carried on a treadmill or in a stationary bicycle.

The post intervention aerobic capacity will be measured at week 3 and 4 with the 6-minute walk test. The main efficacy outcome will be peak oxygen consumption (VO2 peak) and the safety outcomes will be exercise-related adverse events and the program adherence.

This protocol was approved by the Instituto Nacional de Cancerología's Ethical Board

DETAILED DESCRIPTION:
Gastrointestinal - origin cancer is one of the most frequent causes of cancer worldwide ; the primary surgical management is the standard treatment, however, the postoperative complications rate could be up to 35% . Patients with gastrointestinal - origin cancer often experience physical deconditioning; this could lead to an increased risk of complications, especially when they require major abdominal procedures.

It has been suggested that physical training in the preoperative period could improve their condition, reducing the risk of complications. Although this topic has been investigated, it has not been established yet the best short preoperative aerobic exercise program to enhance the aerobic capacity in patients with gastrointestinal cancer who are going to be to surgical primary management, and consequently, to help patients dealing with the physiological stress involved in a surgical intervention.

Main objective:

To determine the efficacy and safety of a 4 weeks preoperative exercise program in patients with gastrointestinal cancer scheduled for primary surgery.

Materials and methods:

This is a Phase II single arm clinical trial that will include patients between 45 and 70 years, with confirmed gastrointestinal cancer (gastric, liver, colon or rectal cancer), scheduled for surgery in 4 weeks or more since recruitment and without electrocardiographic abnormalities.

The patients will be selected from the gastrointestinal unit surgical schedule. The eligible patients will be invited to participate and after their agreement to participate and to do the informed consent process, they will be scheduled to the basal assessment. This aerobic capacity assessment will be done with the 6-minute walk test.

After the basal measurement, two physical therapists will prescribe an individualized aerobic training program in 3 sessions per week during 4 weeks. Each session will last 50 minutes and will be programmed as follows:

* Week 1: heart rate target: 50% of maximum heart rate
* Week 2: heart rate target: 60% of maximum heart rate
* Week 3: heart rate target: 70% of maximum heart rate
* Week 4: heart rate target: 60% of maximum heart rate

The aerobic exercise will be carried on a treadmill or in a stationary bicycle, according to the patient's preferences and will be supervised by a physical therapist.

The post intervention aerobic capacity will be measured at week 3 and 4 with the 6-minute walk test. The main efficacy outcome will be peak oxygen consumption (VO2 peak) and the safety outcomes will be exercise-related adverse events and the program adherence.

This protocol was approved by the Instituto Nacional de Cancerología's Ethical Board.

ELIGIBILITY:
Inclusion criteria:

* 45 to 70 years
* Confirmed diagnosis of gastric, hepatic, colon or rectal cancer.
* Live in Bogota for at least 3 months
* Hemoglobin concentration superior to 10g/dL
* Primary surgery date scheduled in the next 4 weeks or more since eligibility assessment
* ECOG score 0 or 1

Exclusion criteria:

* Behavior or cognitive impairment
* musculoskeletal impairment
* any exercise contraindication (fracture or sprains in the last 2 months, severe osteoarthritis, tendinitis)
* Uncontrolled metabolically comorbidities (diabetes, hypertension, hyperlipidemia)
* Presence of obstructive or restrictive pulmonary disease
* Enrolled in another supervised exercise program
* Major electrocardiographic abnormalities.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen comsumption | 4 weeks after the exercise program beginning
  peak oxygen consumption measured in ml/kg/min using the American College of Sports Medicine's equation

SECONDARY OUTCOMES:
exercise-related adverse events | 3 and 4 weeks after the exercise program beginning
  any unexpected reaction secondary to the exercise program. This could be mild (nausea, fall, joint pain, tendinitis) or severe (syncope, fracture, myocardial infarction).
program adherence | 3 weeks after the exercise program beginning.
  frequency of patients who will complete at least the 3 week program.
Peak oxygen comsumption - 3 weeks | 3 weeks after the exercise program beginning
  peak oxygen consumption measured in ml/kg/min using the American College of Sports

CONTACTS AND LOCATIONS:
Overall Officials: Oscar A Guevara, MD MSc, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto Nacional de Cancerología, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Background] Pardo C, Cendales R. Incidencia, prevalencia y mortalidad de Cáncer en Colombia, 2007-2011: Instituto Nacional de Cancerología; 2015.
- [Background] Chicharro, JL., Vaquero, AF. (2006). Fisiología del ejercicio. Ed. Médica Panamericana.
- [Background] Schmidt K, Vogt L, Thiel C, Jager E, Banzer W. Validity of the six-minute walk test in cancer patients. Int J Sports Med. 2013 Jul;34(7):631-6. doi: 10.1055/s-0032-1323746. Epub 2013 Feb 26. PMID 23444095
- [Result] Veen EJ, Steenbruggen J, Roukema JA. Classifying surgical complications: a critical appraisal. Arch Surg. 2005 Nov;140(11):1078-83. doi: 10.1001/archsurg.140.11.1078. PMID 16301444
- [Result] Worster B, Holmes S. A phenomenological study of the postoperative experiences of patients undergoing surgery for colorectal cancer. Eur J Oncol Nurs. 2009 Dec;13(5):315-22. doi: 10.1016/j.ejon.2009.04.008. Epub 2009 May 30. PMID 19482512
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Martos-Benitez FD, Gutierrez-Noyola A, Echevarria-Victores A. Postoperative complications and clinical outcomes among patients undergoing thoracic and gastrointestinal cancer surgery: A prospective cohort study. Rev Bras Ter Intensiva. 2016 Jan-Mar;28(1):40-8. doi: 10.5935/0103-507X.20160012. PMID 27096675
- [Result] Wilson RJ, Davies S, Yates D, Redman J, Stone M. Impaired functional capacity is associated with all-cause mortality after major elective intra-abdominal surgery. Br J Anaesth. 2010 Sep;105(3):297-303. doi: 10.1093/bja/aeq128. Epub 2010 Jun 23. PMID 20573634
- [Result] Moyes LH, McCaffer CJ, Carter RC, Fullarton GM, Mackay CK, Forshaw MJ. Cardiopulmonary exercise testing as a predictor of complications in oesophagogastric cancer surgery. Ann R Coll Surg Engl. 2013 Mar;95(2):125-30. doi: 10.1308/rcsann.2013.95.2.125. PMID 23484995
- [Result] Jin F, Chung F. Minimizing perioperative adverse events in the elderly. Br J Anaesth. 2001 Oct;87(4):608-24. doi: 10.1093/bja/87.4.608. PMID 11878732
- [Result] Loewen GM, Watson D, Kohman L, Herndon JE 2nd, Shennib H, Kernstine K, Olak J, Mador MJ, Harpole D, Sugarbaker D, Green M; Cancer and Leukemia Group B. Preoperative exercise Vo2 measurement for lung resection candidates: results of Cancer and Leukemia Group B Protocol 9238. J Thorac Oncol. 2007 Jul;2(7):619-25. doi: 10.1097/JTO.0b013e318074bba7. PMID 17607117
- [Result] Jones LW, Liang Y, Pituskin EN, Battaglini CL, Scott JM, Hornsby WE, Haykowsky M. Effect of exercise training on peak oxygen consumption in patients with cancer: a meta-analysis. Oncologist. 2011;16(1):112-20. doi: 10.1634/theoncologist.2010-0197. Epub 2011 Jan 6. PMID 21212429
- [Result] Pouwels S, Stokmans RA, Willigendael EM, Nienhuijs SW, Rosman C, van Ramshorst B, Teijink JA. Preoperative exercise therapy for elective major abdominal surgery: a systematic review. Int J Surg. 2014;12(2):134-40. doi: 10.1016/j.ijsu.2013.11.018. Epub 2013 Dec 8. PMID 24325942
- [Result] Boereboom C, Doleman B, Lund JN, Williams JP. Systematic review of pre-operative exercise in colorectal cancer patients. Tech Coloproctol. 2016 Feb;20(2):81-9. doi: 10.1007/s10151-015-1407-1. Epub 2015 Nov 27. PMID 26614304
- [Result] Dunne DF, Jack S, Jones RP, Jones L, Lythgoe DT, Malik HZ, Poston GJ, Palmer DH, Fenwick SW. Randomized clinical trial of prehabilitation before planned liver resection. Br J Surg. 2016 Apr;103(5):504-12. doi: 10.1002/bjs.10096. Epub 2016 Feb 11. PMID 26864728
- [Result] Ministerio de la Proteccion Social (Colombia). Guía de práctica clínica (GPC) para la detección temprana, el diagnóstico, tratamiento integral, seguimiento y rehabilitación de pacientes con diagnostico de cáncer de colon y recto 2013.
- [Result] Van Cutsem E, Sagaert X, Topal B, Haustermans K, Prenen H. Gastric cancer. Lancet. 2016 Nov 26;388(10060):2654-2664. doi: 10.1016/S0140-6736(16)30354-3. Epub 2016 May 5. PMID 27156933
- [Result] Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O, Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clin Nutr. 2010 Aug;29(4):434-40. doi: 10.1016/j.clnu.2010.01.004. Epub 2010 Jan 29. PMID 20116145
- [Result] Levett DZ, Grocott MP. Cardiopulmonary exercise testing, prehabilitation, and Enhanced Recovery After Surgery (ERAS). Can J Anaesth. 2015 Feb;62(2):131-42. doi: 10.1007/s12630-014-0307-6. Epub 2015 Jan 22. PMID 25608638
- [Result] Gupta R, Gan TJ. Preoperative Nutrition and Prehabilitation. Anesthesiol Clin. 2016 Mar;34(1):143-53. doi: 10.1016/j.anclin.2015.10.012. PMID 26927744
- [Result] Knols R, Aaronson NK, Uebelhart D, Fransen J, Aufdemkampe G. Physical exercise in cancer patients during and after medical treatment: a systematic review of randomized and controlled clinical trials. J Clin Oncol. 2005 Jun 1;23(16):3830-42. doi: 10.1200/JCO.2005.02.148. PMID 15923576
- [Result] Jones LW, Eves ND, Haykowsky M, Freedland SJ, Mackey JR. Exercise intolerance in cancer and the role of exercise therapy to reverse dysfunction. Lancet Oncol. 2009 Jun;10(6):598-605. doi: 10.1016/S1470-2045(09)70031-2. PMID 19482248
- [Result] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Result] Alcalde-Escribano JR-L, P. Acosta,F. Landa, I. Lorenzo,S, Villeta-Plaza RJE. Estudio Delphi para el desarrollo de pautas de indicación de pruebas preoperatorias. Consenso de anestesiólogos y cirujanos. Rev Calidad Asistencial. 2002;17(1):34-42.
- [Result] Wilmore, JH., Costill, DL. (2004). Fisiología del esfuerzo y del deporte. Editorial Paidotribo.
- [Result] Albouaini K, Egred M, Alahmar A, Wright DJ. Cardiopulmonary exercise testing and its application. Postgrad Med J. 2007 Nov;83(985):675-82. doi: 10.1136/hrt.2007.121558. PMID 17989266
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180